CLINICAL TRIAL: NCT05847556
Title: Development and Validation of the Use of Video Games and Virtual Reality to Enable Autonomous Remote Monitoring of OTotoxicity in High-risk Population Groups.
Brief Title: Video Game Hearing Tests for Remote Monitoring of Ototoxicity
Acronym: VAROT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HH7217
Record Dates: First submitted 2023-03-07; First posted 2023-05-06 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Aminoglycoside Toxicity; Aminoglycoside-Induced Hearing Loss; Hearing Loss; Video Games
MeSH Terms: conditions — Hearing Loss | interventions — Noise

STUDY DESIGN:
Intervention Model Description: Pathway 1: pilot study of non-medical device Pathway 2: observational cohort study of medical device Pathway 3: randomised pilot study of non-medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Monitoring of ototoxicity (Experimental): Video game hearing tests will be used to determine if they can effectively monitor changes in hearing function over time remotely.
  Interventions: Other: video game hearing tests
- Tablet-based audiometry validation (No Intervention): Further validation of tablet-based audiometry compared to formal sound-booth audiometry.
- Audio-training - intervention arm (Experimental): Audio-training with video game hearing tests will be used to determine if it can improve spatial hearing perception.
  Interventions: Other: Audio-training
- Audio-training - control arm (No Intervention): No audio-training but video game hearing tests will be used as a comparator arm to identify if audio-training can improve spatial hearing perception.

INTERVENTIONS:
Other: video game hearing tests — Video game hearing tests (as a non-medical device) used to monitor ototoxicity
  Other Names: SSIN-VR; Spatial Speech in Noise-Virtual Reality
  Arms: Monitoring of ototoxicity
Other: Audio-training — Audio-training (as a non-medical device) used to determine if it can improve spatial hearing perception.
  Other Names: SSIN-Loc training; Spatial Speech in Noise and Localisation Training
  Arms: Audio-training - intervention arm

SUMMARY:
The reason for this clinical trial is to test different ways of carrying out hearing tests to be able to detect for hearing loss within the hospital and at home.

Pathway 1:

The goal of this clinical trial is to learn whether video game hearing tests work well to detect hearing loss caused by antibiotics at home in patients with long-term lung infections.

Pathway 2:

The goal of this clinical trial is to compare tablet-based (iPad) hearing tests with formal sound booth hearing tests in patients attending hospital outpatient clinics.

Pathway 3:

The goal of this clinical trial is to learn whether audio-training improves listening to speech in the presence of background noise. Researchers will compare participants receiving audio-training with those who did not receive audio-training. This will test if audio-training can improve participant's everyday listening experiences.

DETAILED DESCRIPTION:
Aminoglycoside antibiotics are widely used in clinical practice to treat life-threatening infections. However, they are associated with ototoxicity leading to hearing loss, tinnitus and vestibular problems.

Mobile devices such as tablet audiometry have recently been validated as a screening tool for hearing loss in an adult cystic fibrosis cohort demonstrating good sensitivity, specificity and positive predictive value when compared to formal sound booth audiometry (Vijayasingam 2020).

Technology from the BEARS project is being adapted to integrate hearing tests within video games and virtual reality software. This technology (Spatial Speech in Noise virtual reality (SSIN-VR) test) will then be used as a tool to perform hearing tests to see if it can detect ototoxicity in adult patients receiving ototoxic agents. The video game-based virtual reality technology (Spatial Speech in Noise and Localisation (SSIN-Loc Training)) will be used to train and potentially improve spatial hearing. This can be done remotely at the convenience of the patient and aims to be an effective way of monitoring hearing autonomously with high usability.

There are 3 pathways within this study:

Pathway 1 (monitoring ototoxicity) is a pilot study to measure the utility and effectiveness of video game-based virtual reality (SSIN-VR) hearing tests as an effective means to monitor hearing loss in patients receiving ototoxic agents. It will be compared with tablet-based audiometry carried out by non-specialist staff, and formal standard sound-booth extended high-frequency audiometry performed by an audiologist. 30 patients receiving an ototoxic agent, presenting at one of the recruiting centres, will be recruited into this pathway.

Pathway 2 is a prospective observational cohort study which continues to validate the use of tablet-based audiometry compared with formal standard sound-booth extended high-frequency audiometry performed by an audiologist. 80 patients, presenting at one of the recruiting centres, will be prospectively recruited into this pathway.

Pathway 3 is a pilot study which assesses whether audio-training (SSIN-Loc training) with video game-based virtual reality (SSIN-VR) hearing tests can improve spatial hearing perception and speech intelligibility. 30 participants will be recruited into this pathway. They will be randomised to either the intervention group (Arm 1) or the control group (Arm 2). All participants will carry out a baseline video game-based virtual reality hearing (SSIN-VR) test in the first week.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥16 years old intended to receive >1 day of an ototoxic agent (Pathway 1)
* All patients ≥16 years old (Pathways 2 and 3)
* Able to provide informed consent to participate in study (written and witnessed).

Exclusion Criteria:

* Inability of patient to provide informed consent.
* Patients with previous diagnosed visual impairment that cannot be corrected with glasses.
* Inability to attend audiology appointments due to state of health.
* Pregnant women.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Pure-tone thresholds analysed through tablet-based audiometry and standard extended high-frequency audiometry. | For the 4 months that patient is enrolled

SECONDARY OUTCOMES:
Analysis of spatial speech in noise scores from video game-based virtual reality hearing tests. | For the 4 months that patient is enrolled
Interclass correlation coefficient (ICC) with a 95% confidence interval will be used as a measure of reliability. | For the 4 months that patient is enrolled
Sensitivity, specificity and negative predictive value will be analysed to determine utility of video game-based virtual reality and tablet-based audiometry. | For the 4 months that patient is enrolled
Logistical regression modelling to determine risk factors for developing hearing loss | For the 4 months that patient is enrolled
7-point Likert scale questionnaires will be used to evaluate patient satisfaction of video game-based virtual reality hearing tests, audio-training, tablet-based and formal audiometry. | For the 4 months that patient is enrolled
  Attractiveness, perspicuity, efficiency, dependability, simulation and novelty will be interpreted and scaled from -3 (minimum) to +3 (maximum). Scores above +1 indicate a positive impression and values below -1, a negative impression.
Pearsons correlation will be used to identify if demographic variables have an effect on questionnaire results. | For the 4 months that patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Anand Shah, Principal Investigator — Imperial College London; Francis Drobniewski, Study Chair — Imperial College London
Locations (2):
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust, London
  - University Hospitals Dorset NHS Foundation Trust, Poole

REFERENCES:
- [Background] Vijayasingam A, Frost E, Wilkins J, Gillen L, Premachandra P, Mclaren K, Gilmartin D, Picinali L, Vidal-Diez A, Borsci S, Ni MZ, Tang WY, Morris-Rosendahl D, Harcourt J, Elston C, Simmonds NJ, Shah A. Tablet and web-based audiometry to screen for hearing loss in adults with cystic fibrosis. Thorax. 2020 Aug;75(8):632-639. doi: 10.1136/thoraxjnl-2019-214177. Epub 2020 May 14. PMID 32409613
- [Derived] Cheong J, Lowe E, Lee CW, Barbosa C, Gillen L, King E, Premachandra P, Shah A, Drobniewski F. Globally applicable solution to hearing loss screening: a diagnostic accuracy study of tablet-based audiometry. BMJ Open. 2025 May 22;15(5):e097550. doi: 10.1136/bmjopen-2024-097550. PMID 40404318